CLINICAL TRIAL: NCT02639923
Title: The Clinical Relevance of Micro RNAs in Mild Traumatic Brain Injury A Pilot Study
Brief Title: The Clinical Relevance of Micro RNAs in Mild Traumatic Brain Injury
Acronym: mRNA
Status: Completed | Type: Observational
Sponsor: Harald Wolf, MD (Other)
Collaborators: Medical Scientific Fund of the Mayor of Vienna (Other)
Responsible Party: Sponsor-Investigator, Harald Wolf, MD, Oberarzt Dr. Harald Wolf, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: Wolf-7
Record Dates: First submitted 2015-12-02; First posted 2015-12-28 (Estimated); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Brain Injuries, Traumatic
Keywords: TBI; microRNA; S-100B
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 7ml serum are drawn from peripheral blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Minor head injury CCT pos. group: Tbi patients with acute lesion on early cranial computed tomography. Patients consent to have 7ml peripheral blood to be drawn.
  Interventions: Procedure: Drawing of 7ml peripheral blood
- Minor head injury CCT neg. group: Tbi patients without acute lesion on early cranial computed tomography. Patients consent to have 7ml peripheral blood to be drawn.
  Interventions: Procedure: Drawing of 7ml peripheral blood
- Control Group (healthy volunteers): Volunteers without history, signs or symptoms of acute traumatic injuries. Volunteers consent to have 7ml peripheral blood to be drawn.
  Interventions: Procedure: Drawing of 7ml peripheral blood

INTERVENTIONS:
Procedure: Drawing of 7ml peripheral blood — puncture peripheral vein
  Other Names: 7ml serum

SUMMARY:
The aim of this study is to investigate the early serum measurement (<6h after injury) of mRNA miR Let-7i, miR-16 and miR-92 in patients with MHI and intracranial traumatic lesions (CCT pos.) as compared to those in patients with MHI without intracranial traumatic lesions (CCT neg.).

S100B serum levels will be measured in both groups. The usual risk factors for the occurrence of an intracranial hematoma (diagnostic algorithm) will be recorded. Additionally, a group of healthy individuals will serve as a control group.

DETAILED DESCRIPTION:
Patients and Methods

The investigators plan to include 60 patients with minor head injury (MHI) admitted to our hospital within one year (1-2 each week):

1. 30 patients in the CCT pos. group, i.e. patients with an intracranial hematoma on emergency CT scan. 2. 30 patients with MHI in the CCT neg. group, i.e. patients without an intracranial traumatic lesion on emergency CT-scan. 3. Additionally, 30 healthy volunteers will be included.

Patients with multiple injuries i.e. polytraumatized patients, patients with severe traumatic brain injury, patients with open fractures and fractures of the long bones, as well as pregnant patients and patients <18 years, are excluded from the study.

Patients with a GCS (Glascow Coma Scale) of 13-15 are usually able to consent to be enrolled in the clinical trial. Generally, their reasoning and judgment is not impaired.

The objective of the study is to compare 3 groups on the microRNA serum levels.

The investigators plan to draw blood from a peripheral catheter in the patients of groups 1 and 2 (within 6 hours) after arrival at the hospital together with the routine laboratory investigations. Additionally, blood will be obtained from healthy volunteers (group 3).

ELIGIBILITY:
Inclusion Criteria:

* TBI with GCS 13-15

Exclusion Criteria:

* Patients with multiple injuries i.e. polytraumatized patients, patients with severe traumatic brain injury, patients with open fractures and fractures of the long bones, as well as pregnant patients and patients <18 years, are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to include 60 patients with minor head injury (MHI) GCS 13-15 admitted to our hospital within one year (1-2 each week).
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2016-01; Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Hypothesis: Significant elevation or decrease of the mRNAs miR Let-7i, miR-16 and miR-92 among the study groups | 6 hours
  non of the measured biomarker shows a significant difference between the 3 study groups

CONTACTS AND LOCATIONS:
Overall Officials: Harald Wolf, M.D., Principal Investigator — Department for Trauma Surgery, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Result] Balakathiresan N, Bhomia M, Chandran R, Chavko M, McCarron RM, Maheshwari RK. MicroRNA let-7i is a promising serum biomarker for blast-induced traumatic brain injury. J Neurotrauma. 2012 May 1;29(7):1379-87. doi: 10.1089/neu.2011.2146. Epub 2012 Apr 13. PMID 22352906
- [Result] Sharma A, Chandran R, Barry ES, Bhomia M, Hutchison MA, Balakathiresan NS, Grunberg NE, Maheshwari RK. Identification of serum microRNA signatures for diagnosis of mild traumatic brain injury in a closed head injury model. PLoS One. 2014 Nov 7;9(11):e112019. doi: 10.1371/journal.pone.0112019. eCollection 2014. PMID 25379886
- [Result] Redell JB, Moore AN, Ward NH 3rd, Hergenroeder GW, Dash PK. Human traumatic brain injury alters plasma microRNA levels. J Neurotrauma. 2010 Dec;27(12):2147-56. doi: 10.1089/neu.2010.1481. Epub 2010 Nov 23. PMID 20883153
- [Result] Redell JB, Zhao J, Dash PK. Altered expression of miRNA-21 and its targets in the hippocampus after traumatic brain injury. J Neurosci Res. 2011 Feb;89(2):212-21. doi: 10.1002/jnr.22539. Epub 2010 Dec 8. PMID 21162128